CLINICAL TRIAL: NCT03141229
Title: Gesundheit, Integration, Konzentration: Achtsamkeitsbasierte Stabilisierung Von LehrerInnen Und SchülerInnen
Brief Title: Health, Integration, Concentration: Mindfulness in Schools
Acronym: GIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Ministerium für Schule und Weiterbildung, Land Nordrhein-Westfalen (Unknown); Ministerium für Gesundheit, Emanzipation, Pflege und Alter, Land Nordrhein-Westfalen (Unknown)
Responsible Party: Principal Investigator, Holger Cramer, Director of research, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-6998-BO
Record Dates: First submitted 2017-02-09; First posted 2017-05-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Mindfulness; Child Development; Burnout Syndrome
Keywords: MBSR; Children; Teacher; School; Burnout; Classroom behavior
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Note: Either teacher and pupils are included in this study. We anticipate a number of 100 teacher and 500 pupils participating. Data from teacher and pupils will be analyzed separately.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): One school semester MBSR training for teacher; followed by one school semester mindfulness training for children and one school semester follow-up period.
  Interventions: Behavioral: Mindfulness based stress reduction
- Waitlist (Other): One school semester waitlist; followed by one school semester MBSR training for teacher and one school semester MBSR training for children.
  Interventions: Behavioral: Mindfulness based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness based stress reduction
  Other Names: MBSR

SUMMARY:
Mindfulness training for teacher and children of primary schools. Blinded and controlled study design. Burnout as primary outcome for teacher and classroom behavior for children.

ELIGIBILITY:
Inclusion Criteria:

* reading ability
* positive declaration of consent

Exclusion Criteria:

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12; Primary Completion 2018-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Burnout (Teacher) assessed with the Burnout-Screening-Scale | Baseline; Timepoint 1 (4 month); Timepoint 2 (12 month); Timepoint 3 (16 month)
  Burnout-Screening-Scale (Change from baseline)
Classroom climate pupils | Baseline; Timepoint 1 (4 month); Timepoint 2 (12 month); Timepoint 3 (16 month)
  Emotional and social school experience questionnaire (Change from baseline)

SECONDARY OUTCOMES:
Stress and Anxiety (Teacher) assessed with the Stress and Anxiety Inventory | Baseline; Timepoint 1 (4 month); Timepoint 2 (12 month); Timepoint 3 (16 month)
  Stress and Anxiety Inventory for teacher (Change from baseline)
Mindfulness (Teacher) assessed with the Freiburg Mindfulness Inventory | Baseline; Timepoint 1 (4 month); Timepoint 2 (12 month); Timepoint 3 (16 month)
  Freiburg Mindfulness Inventory (Change from baseline)
Concentration (pupils) assessed with a d2-Concentration assessment tool | Baseline; Timepoint 1 (4 month); Timepoint 2 (12 month); Timepoint 3 (16 month)
  d2-Concentration assessment tool (Change from baseline)
Health-related Quality of Life (pupils) assessed with the Kidscreen-10 | Baseline; Timepoint 1 (4 month); Timepoint 2 (12 month); Timepoint 3 (16 month)
  Kidscreen-10 (Change from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, MD, Principal Investigator — Universität Duisburg-Essen, Medizinische Fakultät, Klinik für Naturheilkunde und Integrative Medizin
Locations (1):
- Schulamt Stadt Solingen, Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No